CLINICAL TRIAL: NCT02658123
Title: Reducing Readmissions in High-Risk Ostomates
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decline in enrollment, lack of efficacy, and completion of funding accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201601014
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Ileostomy
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Standard of care (Active Comparator): * Standard of care pre-operative education
  * Standard of care home health visits
  * Standard of care follow-up post-operative visits with surgeon and CWOCN
  * At 30-days post hospital discharge, the participant will:
    * See the physician
    * Turn in Patient Data Collection Form
    * Turn in Healthcare Utilization Form
    * Complete The City of Hope QOL Survey for Ostomy Patients
    * Ostomy assessment with a CWOCN, including photo of ostomy site
  Interventions: Other: Pre-operative education (standard of care); Other: Home health care visits (standard of care); Other: Follow-up post-operative visits; Other: Patient Data Collection Form; Other: Healthcare Utilization Form; Other: The City of Hope QOL Survey for Ostomy Patients
- Group B: Phone call (Experimental): * Standard of care pre-operative education
  * Standard of care home health visits
  * Standard of care follow-up post-operative visits with surgeon and CWOCN
  * Telephone call 48-72 hours post-discharge from CWOCN/PA to evaluate tolerability to foods/fluids, activity level, screen for red-flags, review/assess for medication, reviewing pouching of ostomy, review patient's ability to obtain supplies, provide continued education, discuss proper use of durable medical equipment/frequency of pouch changes, and complete Patient Assessment Form.
  * At 30-days post hospital discharge, the participant will:
    * See the physician
    * Turn in Patient Data Collection Form
    * Turn in Healthcare Utilization Form
    * Complete The City of Hope QOL Survey for Ostomy Patients
    * Ostomy assessment with a CWOCN, including photo of ostomy site
  Interventions: Other: Pre-operative education (standard of care); Other: Home health care visits (standard of care); Other: Follow-up post-operative visits; Other: Patient Data Collection Form; Other: Healthcare Utilization Form; Other: The City of Hope QOL Survey for Ostomy Patients; Other: Phone call with CWOCN or PA

INTERVENTIONS:
Other: Pre-operative education (standard of care)
Other: Home health care visits (standard of care)
Other: Follow-up post-operative visits
Other: Patient Data Collection Form — -Form that contains date, area to record number of pouches, and if home health care visit took place.
Other: Healthcare Utilization Form — * Form for patient to record if they visited an emergency room or urgent care or if they were hospitalized
  * Form allows patient to record reason for visit and date of visit
Other: The City of Hope QOL Survey for Ostomy Patients — * Consists of 47 questions asking various physical, psychological, sexual, work-related, and demographic questions.
  * Additional 34 questions on how the ostomy affects quality of life. Answers range from 0=not at all to 10=severe problem.
Other: Phone call with CWOCN or PA
  Arms: Group B: Phone call

SUMMARY:
Preventing complications and readmission after ostomy surgery will decrease the cost of healthcare, improve patient safety, reduce the cost of durable medical equipment required by ostomates, ensure continued specialized care is available, and potentially improve both short and long-term quality of life (QOL) for patients by reducing morbidity and mortality associated with ostomy surgery. The purpose of this study is to measure the effectiveness of patient centered interventions/care pathways and to determine the impact on healthcare utilization, 30-day hospital readmissions, and QOL.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo surgery that will result in the creation of an ileostomy.
* Agreed to receive home healthcare.
* At least 18 years of age.
* Speaks English.
* Has access to telephone.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

-Unwilling or unable to receive home health care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Impact of early implementation of post-operative assessment by Certified Wound Ostomy Continence Nurse (CWOCN) or physician's assistant (PA) via follow-up telephone call on health care utilization as measured by number of emergency room visits | Within the first 30 days after hospital charge (up to approximately 37 days)
Impact of early implementation of post-operative assessment by CWOCN or PA via follow-up telephone call on health care utilization as measured by number of hospitalizations | Within the first 30 days after hospital charge (up to approximately 37 days)
Impact of early implementation of post-operative assessment by CWOCN or PA via follow-up telephone call on health care utilization as measured by number of urgent care visits | Within the first 30 days after hospital charge (up to approximately 37 days)

SECONDARY OUTCOMES:
Impact that the early telephone follow-up and evaluation have on the number of office visits | First 30 days after hospital discharge (approximately 37-52 days after admission)
impact that the early telephone follow-up and evaluation have on the number of phone calls to the office | First 30 days after hospital discharge (approximately 37-52 days after admission)
Impact that the early telephone follow-up and evaluation have on durable medical equipment (DME) usage | 30-day CWOCN visit (approximately 37-52 days after admission)
Impact that the early telephone follow-up and evaluation have on peristomal skin irritation DET score | 30-day CWOCN visit (approximately 37-52 days after admission)
  -PeriPeristomal Skin Assessment/DET score based on discoloration, severity of discoloration, erosion, severity of erosion, tissue overgrowth, and severity of tissue overgrowth
Impact that the early telephone follow-up and evaluation have on the scores of QOL (quality of life) questionnaire | 30-day clinical visit (approximately 37-52 days after admission)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Hunt, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu